CLINICAL TRIAL: NCT07254676
Title: Effects of Virtual Reality-Enhanced Rehabilitation on Upper Limb Recovery in Acute Post-Stroke Patients: a Pilot Study
Brief Title: Virtual Reality-Enhanced Rehabilitation for Upper Limb Recovery in Acute Post-Stroke Patients
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Tadeja Hernja Rumpf, Principal Investigator, University Medical Centre Maribor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UKC-MB-KME-36/21; IRP-2021/02-08 (Other Grant/Funding Number: UKC Maribor)
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Acute Stroke Intervention; Rehabilitation Exercise
Keywords: virtual reality; stroke rehabilitation; upper limb; cognition; acute phase
MeSH Terms: interventions — Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to the experimental group (VR training in addition to CRT) or the control group (only CRT) using sealed envelopes with group tasks in numerical sequence.
Who Masked: Investigator
Masking Description: Therapists who will evaluate participants with scales will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR + CRT (Virtual reality-enhanced rehabilitation plus Conventional rehabilitation therapy) (Experimental): The experimental group will receive physiotherapy and occupational therapy (manual therapy techniques, passive and active-assisted mobilisation, scapular mobilisation, and task-specific training such as horizontally moving an object across a surface), ten sessions over two weeks of 60 minutes per session and an additional 15 minutes of virtual-reality (VR) training per session using the Bimeo PRO system (Kinestica d.o.o., Slovenia) in a unimanual, two-dimensional configuration on a flat surface, with continuous therapist supervision.
  Interventions: Behavioral: Virtual Reality-enhanced rehabilitation; Other: Conventional rehabilitation therapy (CRT)
- CRT (Conventional rehabilitation therapy) (Active Comparator): The control group will receive ten sessions over two weeks of physiotherapy and occupational therapy (manual therapy techniques, passive and active-assisted mobilisation, scapular mobilisation, and task-specific training such as horizontally moving an object across a surface), 60 minutes per session.
  Interventions: Other: Conventional rehabilitation therapy (CRT)

INTERVENTIONS:
Behavioral: Virtual Reality-enhanced rehabilitation — Dose of practice and difficulty:
  In each VR session, participants will perform three tasks, completing one trial of each-reaching, tracking, and labyrinth-with no within-session repetitions. Across ten sessions, participants will complete ten trials of each task (30 trials in total). Task difficulty will be fixed and identical for all participants throughout the intervention (no automatic progression or therapist-driven difficulty changes).
  Adherence, tolerability, and adverse events:
  Participants will be scheduled to complete the prescribed VR dose (10 sessions; 150 minutes total). Adherence will be recorded at each session. Serious adverse events are not expected; all adverse events will be actively monitored and documented.
  Arms: VR + CRT (Virtual reality-enhanced rehabilitation plus Conventional rehabilitation therapy)
Other: Conventional rehabilitation therapy (CRT) — Physiotherapy and occupational therapy: manual therapy techniques, passive and active-assisted mobilisation, scapular mobilisation, and task-specific training such as horizontally moving an object across a surface), 60 minutes per session.
  Other Names: physiotherapy; occupational therapy

SUMMARY:
Post-stroke rehabilitation is essential for maximising motor recovery. Virtual reality (VR) is emerging as a promising adjunct to conventional therapy (CRT), potentially enhancing upper limb motor outcomes. The goals of the study are:

1. To evaluate the efficiency of VR in addition to CRT on upper limb function in the acute phase of post-stroke rehabilitation, which is underrepresented in the literature.
2. To explore the relationship between cognitive impairment and upper limb motor recovery using VR.

The investigators hypothesise that combining VR and CRT improves upper limb functional outcomes in acute stroke beyond the effects of CRT.

DETAILED DESCRIPTION:
The investigators will conduct a prospective randomised single- blind pilot controlled trial to evaluate the efficacy of VR-based rehabilitation with the Bimeo PRO system in improving upper limb function in acute post-stroke patients. Participants will be randomly assigned to a two-week program of VR training combined with conventional therapy (experimental group) or conventional therapy alone (control group).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* First-ever acute stroke, occurring <7 days before therapy start.
* Upper-limb activity limitation with some preserved function (e.g., ability to grasp).
* Able to understand instructions and provide informed consent.

Exclusion Criteria:

* Severe cognitive impairment that precludes following instructions.
* Aphasia or severe visual/hearing impairment that prevents meaningful participation.
* End-stage/terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
The Fugl-Meyer Upper Extremity Assessment (FMA-UE) | Change from baseline to 2 weeks (end of intervention)
  Fugl-Meyer Upper Extremity Assessment (FMA-UE). Will evaluate post-stroke body functions-motor function, sensation, passive joint motion, and joint pain. Scoring will sum all item scores to a total of 0-126, with higher scores indicating better function.
The Wolf Motor Function Test (WMFT) | Change from baseline to 2 weeks (end of intervention)
  Wolf Motor Function Test (WMFT). Will assess upper-limb performance with 17 items (2 strength items and 15 timed tasks) that progress from proximal to distal/whole-limb movements. Outcomes will include task times and the Functional Ability Scale (FAS); the mean FAS will be computed as total FAS/15 (range 0-5).
Grip strength | Change from baseline to 2 weeks (end of intervention)
  Grip strength. Will be measured in kilograms using a calibrated hand dynamometer. Participants will perform three maximal efforts with the affected hand while seated (elbow 90°, forearm neutral); the best of three will be recorded for analysis.

SECONDARY OUTCOMES:
The National Institutes of Health Stroke Scale (NIHSS) | Change from baseline to 2 weeks (end of intervention)
  The NIHSS is a comprehensive assessment tool used to evaluate the severity of a stroke. The scale generates scores ranging from 0, denoting the absence of deficits, to 46, signifying severe impairment.
The Modified Rankin Scale (mRS) | Change from baseline to 2 weeks (end of intervention)
  The Modified Rankin Scale (mRS) is a widely utilised and reliable functional assessment tool in clinical trials for stroke patients. Deviating from task-specific evaluations, the mRS measures the level of independence on a scale of 0 to 6.
The Montreal Cognitive Assessment (MoCA) | Change from baseline to 2 weeks (end of intervention)
  The Montreal Cognitive Assessment (MoCA) serves as a cognitive screening instrument, encompassing the evaluation of visuospatial/executive function, naming, memory, attention, language, abstraction, recall, and orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Tadeja Hernja Rumpf, MD, PhD, Principal Investigator — University Medical Centre Maribor, Ljubljanska 5, 2000 Maribor, Slovenia
Locations (1):
- University Medical Centre Maribor, Ljubljanska 5 Maribor, Slovenia, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to small sample size and increased re-identification risk under GDPR. Aggregate results, study protocol, and statistical analysis plan will be made available upon publication.

REFERENCES:
- [Background] Karamians R, Proffitt R, Kline D, Gauthier LV. Effectiveness of Virtual Reality- and Gaming-Based Interventions for Upper Extremity Rehabilitation Poststroke: A Meta-analysis. Arch Phys Med Rehabil. 2020 May;101(5):885-896. doi: 10.1016/j.apmr.2019.10.195. Epub 2019 Dec 7. PMID 31821799
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493
- [Background] Chen X, Liu F, Lin S, Yu L, Lin R. Effects of Virtual Reality Rehabilitation Training on Cognitive Function and Activities of Daily Living of Patients With Poststroke Cognitive Impairment: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2022 Jul;103(7):1422-1435. doi: 10.1016/j.apmr.2022.03.012. Epub 2022 Apr 10. PMID 35417757
- [Background] Li J, Wang J, Wu B, Xu H, Wu X, Zhou L, Deng B. Association Between Early Cognitive Impairment and Midterm Functional Outcomes Among Chinese Acute Ischemic Stroke Patients: A Longitudinal Study. Front Neurol. 2020 Feb 26;11:20. doi: 10.3389/fneur.2020.00020. eCollection 2020. PMID 32174878
- [Background] Kim WS, Cho S, Ku J, Kim Y, Lee K, Hwang HJ, Paik NJ. Clinical Application of Virtual Reality for Upper Limb Motor Rehabilitation in Stroke: Review of Technologies and Clinical Evidence. J Clin Med. 2020 Oct 21;9(10):3369. doi: 10.3390/jcm9103369. PMID 33096678
- [Background] Gorsic M, Cikajlo I, Novak D. Competitive and cooperative arm rehabilitation games played by a patient and unimpaired person: effects on motivation and exercise intensity. J Neuroeng Rehabil. 2017 Mar 23;14(1):23. doi: 10.1186/s12984-017-0231-4. PMID 28330504
- See also: research projects — https://www.ukc-mb.si